CLINICAL TRIAL: NCT01673945
Title: Forward Viewing US Endoscope Versus Standard Viewing US Endoscope in the Performance of EUS-guided Fine Needle Aspiration of Solid Lesions of the Gastrointestinal Tract and of Adjacent Organs: A Prospective Randomized Controlled Study
Brief Title: FV-EUS Endoscope Versus CLA-EUS for EUS-FNA of Solid Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: University of Amsterdam (Other); Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Guido Costamagna, Professor of Surgery, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: P69/CE/2011
Record Dates: First submitted 2012-07-12; First posted 2012-08-28 (Estimated); Last update posted 2019-07-26 (Actual); Status verified 2019-07

CONDITIONS: Solid Lesions of the GI Tract or of Adjacent Organs
Keywords: EUS-FNA, Forward viewing EUS scope, Curvilinear EUS scope
MeSH Terms: interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- EUS-FNA with the CLA-EUS (Active Comparator): patients examined with the CLA-EUS
  Interventions: Device: EUS-guided fine needle aspiration
- EUS-FNA With the FV-EUS (Experimental): patients examined with the FV-EUS
  Interventions: Device: EUS-guided fine needle aspiration

INTERVENTIONS:
Device: EUS-guided fine needle aspiration — Each patient will undergo examination with the CLA-EUS or the FV-EUS, which will be selected based on the randomization process. FV-EUS will be performed using the newly available FV -EUS scope (TGF-Y0001-UC) that is compatible with last generation Aloka alpha 10. First, search of the presumed lesion will be performed and once visualize, its characteristics (size, echogenicity, margins, etc) will be recorded on data collection sheet. Fine needle aspiration will be performed under EUS guidance using a 19- ,22- or a 25-gauge fine needle or procore needles depending on endoscopist's preference

SUMMARY:
The intent of this study is to compare the performance of the CLA-EUS versus the FV-EUS in the performance of EUS-FNA of patients with solid lesions of the GI tract and of adjacent organs, with the aim of establishing for which lesions and from which location the capability of the FV-EUS will be superior, equal or, inferior to the CLA-EUS

DETAILED DESCRIPTION:
Recently, a forward viewing linear echoendoscope (FV-EUS) has been developed with the aim of potentially expanding the therapeutic applications of EUS. This prototype is a modification of the CLA scope and it is characterized primarily by a shifting of the orientation of the endoscopic and US views from oblique to forward. The US transducer is located adjacent to the working channel, at the endoscope tip, to display a forward-viewing image along to a scanning plane that is parallel to the insertion direction with a 90° scanning range. It has a 3.7 mm working channel without elevator, which allows exit of the FNA needle or any other accessory used parallel to the longitudinal axis of the scope.

Preliminary experiences with this scope have reported potential advantages over the conventional linear scope (CLA-EUS) for pseudocysts drainage and for hilar biliary strictures. Moreover, a large experience still unpublished from the Catholic University, Rome, Italy in the use of the FV-EUS for FNA of solid and cystic lesions throughout the GI tract has shown the FV-EUS to be highly effective with a performance that seems at least comparable to that of the CLA-EUS. To date, however, no data comparing the performance of both scopes for FNA of target lesions are available to better clarify the advantages and disadvantages of one scope over the other.

We designed a randomized comparative trial in which patients will be randomized to undergo examination with CLA-EUS or with FV-EUS. In case of failure of: (i) visualization of the presumed lesion; (ii) failure in performing the FNA with the scope used based on randomization, a second attempt will be made using the other scope.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of a solid lesion in the GI tract or in one of the adjacent organs identified at abdominal US, CT, MRI/MRCP that needs to be samples with EUS-FNA because unresectable or because tissue characterization is needed to decide further treatment modalities
2. Age greater than 18.
3. Absence of histological or cytological confirmation of malignancy.
4. Informed consent obtained.

Exclusion Criteria:

1. Patients with active coagulopathy that cannot be corrected after administration of plasma.
2. Resectable lesions that does not need tissue characterization to decide treatment modalities.
3. Pregnancy.
4. Patients who cannot give inform consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2012-06; Primary Completion 2014-07 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Technical performance of the CLA-EUS versus FV-EUS for EUS-FNA | 6 months
  (i)Successful lesion identification. (ii)Successful execution of EUS-FNA proved by EUS image confirming the needle into the lesion.

SECONDARY OUTCOMES:
Diagnostic performance of the CLA-EUS versus FV-EUS for EUS-FNA | 6 months
  sensitivity, specificity, and diagnostic accuracy of EUS-FNA performed with the two different EUS scopes in the evaluation of solid lesions will be determined and compared
Ease of procedure | 6 months
  Ease of the procedure will be graded on a analog 5 point score as listed in the table below.
  Physician will be asked to answer the following questions:
  * Ease of visualization?
  * Ease of puncturing?
  * Ease of moving back and forth inside the lesion?
  * Ease of overall procedure?
Rate of complications | 1 month
  Rate of bleeding, pancreatitis, infection and perforation for each procedure will be measured by observation of the patient in the recovery area soonafter and one hour after completion of the procedure. The rate of pancreatitis and infection rate will be also assessed at 24 hours by visiting or calling the patients if discharged

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Larghi, MD, Principal Investigator — Universita' del Sacro Cuore
Locations (3):
- Erasme University Hospital, Brussels, Belgium
- Universita' del Sacro Cuore, Rome, Italy
- University of Amsterdam medical center, Amsterdam, Netherlands

REFERENCES:
- [Derived] Larghi A, Ibrahim M, Fuccio L, Lekkerkerker S, Eisendrath P, Frazzoni L, Fockens P, La Marca M, van Hooft JE, Deviere J, Costamagna G. Forward-viewing echoendoscope versus standard echoendoscope for endoscopic ultrasound-guided tissue acquisition of solid lesions: a randomized, multicenter study. Endoscopy. 2019 May;51(5):444-451. doi: 10.1055/a-0790-8342. Epub 2018 Nov 29. PMID 30497087